CLINICAL TRIAL: NCT03689530
Title: UPSTART: Using Peer Support to Aid in Prevention and Treatment in Prediabetes
Brief Title: Using Peer Support to Aid in Prevention and Treatment in Prediabetes
Acronym: UPSTART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Kaiser Foundation Research Institute (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mary Ellen Michele Heisler, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00135745; 1R18DK113403-01 (NIH)
Record Dates: First submitted 2018-09-24; First posted 2018-09-28 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: PreDiabetes
Keywords: peer support
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Support Arm. (Experimental): Participants randomized to peer support will be matched with a peer supporter.
  Interventions: Behavioral: Peer Support
- Enhanced Usual Care (Active Comparator): Participants randomized to enhanced usual care will receive brief education and folder of information and resources.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Peer Support — Participants will be paired with a peer supporter. They will meet in person one time and then be in contact by phone or texting on a weekly basis for the first 6 months of a year.
  During the final six months of the year, the peer supporter and participant will be in touch at least monthly. The peer supporter will help link participants to existing health system and community diabetes prevention programs, support their engagement in formal programs, maintain achieved gains, and support participants to initiate and sustain healthy behaviors to prevent diabetes.
  The 95 peer supporters who consented to participate in the study are included in this arm, along with the participants who were randomized to this arm, in the participant flow. The peer supporters were not randomized to the arm; rather, they consented to deliver the intervention. Although 95 consented, only 68 met with at least one peer, the first step in intervention delivery.
  Arms: Peer Support Arm.
Behavioral: Enhanced Usual Care — Participants will receive brief education and folder of information and resources.
  Arms: Enhanced Usual Care

SUMMARY:
An estimated 86 million adults in the United States have prediabetes, and low-income Latino and African American adults have disproportionately high rates compared to non-Hispanic adults. Structured lifestyle interventions can prevent or delay type 2 diabetes in these at-risk populations and now are widely offered at community organizations and health systems. Yet, uptake of and engagement in available formal programs is very low. Low-income adults in particular face multiple barriers to navigating, engaging in, and sustaining involvement in available programs and lifestyle behaviors found to decrease progression to diabetes. It is critically important to develop and evaluate innovative approaches to increase uptake, engagement, and maintenance of gains in diabetes prevention activities. Peer support has been shown in the investigators' and others' effectiveness trials to be a sustainable, effective approach for positive behavior change and improved outcomes in adults with diabetes and other chronic conditions. The study team's pilot work suggests such approaches are feasible and acceptable among low-income Latino and African American patients with prediabetes to prevent chronic disease and better navigate their health care systems to obtain healthy lifestyle counseling and support. However, such peer support models among Latino, African American, and other low-income adults with prediabetes have not yet been rigorously evaluated. Accordingly, the study will conduct a parallel, two-arm randomized controlled trial in primary care centers in two different health systems that serve multi-ethnic communities with a high concentration of Latinos and African Americans and diverse socio-economic backgrounds. The study will compare enhanced usual care (providing referrals to diabetes prevention programs and resources) with a model of a structured behavioral change intervention supplementing enhanced referral to programs and resources with peer support to help link adults with prediabetes to existing health system and community diabetes prevention programs, to support their engagement in formal programs, maintain achieved gains, and support participants to initiate and sustain healthy behaviors to prevent diabetes.

DETAILED DESCRIPTION:
The intervention seeks to address the need to test in routine primary care evidence-based approaches to increase uptake, engagement, and maintenance of healthy behaviors necessary to decrease progression to diabetes among primary care patients with prediabetes, especially low-income and racial and ethnic minority adults with prediabetes. The study will conduct a parallel, two-armed, randomized controlled pragmatic clinical trial including adults with prediabetes at two primary care centers in two different health systems: Kaiser Permanente Northern California and the University of Michigan Health System. Each health system received IRB approval from its own IRB to accommodate site-specific nuances in its implementation. The trial will evaluate whether adding a 12-month predominantly telephone-based volunteer peer support program (UPSTART) to health care provider counseling and referral to diabetes prevention programs leads to greater improvements in A1c, the weight loss, and waist circumference than health care provider counseling and referral alone (Aim 1). The study will also compare differences in reported physical activity, diet, and enrollment and engagement in diabetes prevention programs as potential mediators as well as autonomous motivation, behavior-specific self-efficacy, patient activation, and perceived support; and moderators such as health literacy (Aim 2). To enhance adoption of the intervention by the two study health systems and dissemination to other health systems if effective, the study will evaluate costs and use an integrated RE-AIM and Consolidated Framework for Implementation Research (CFIR) framework to evaluate processes of intervention implementation in the two primary care settings (Aim 3). The study duration will be 5 years, to allow for peer supporter and patient recruitment, completion of the 12-month program, and assessment of outcomes at 6 months and at 12 months.

The study will use mixed methods-i.e., the collection, analysis, and combining of both quantitative and qualitative data-to investigate elements important for implementation and dissemination. The study will gather data on how peer supporters, primary care clinic staff, and patients experience the intervention and how the experiences of participants together with the trial's results suggest the study should modify the intervention. Using this approach, the study aim to ensure that the intervention has the greatest possible likelihood of adoption in both UMHS and KPNC health systems should the study find it has positive effects on processes and outcomes of care. The UPSTART intervention is designed for peers to interact and provide support in a way that is autonomy supportive with the goal of enhancing autonomous motivation and self-efficacy for healthy behaviors. The study will hold periodic initial trainings for new peer supporters over the study period. In addition, peer supporters will receive: 1) routine, structured check-ins that will include monthly peer support group meetings (with option to call in) to allow exchange; 2) back-up support: offering peer supporters contact information for staff who they can call; and 3) continuing education and booster training at the monthly group meetings to enrich their skill sets and knowledge.

The peer supporters were included in the total number of participant numbers for the trial and in the intervention arm in the study flow portion of this record because they were consented. Demographic characteristics of the peer supporters are also reported. However, they were not randomized; they were recruited to deliver the intervention to recruited participants with prediabetes whose outcomes we aimed to improve through the delivered intervention. The peer supporters' involvement was to deliver the intervention to the participants who were randomized to either receive the peer support intervention or to enhanced usual care. The study consented the peer supporters because they completed surveys at three time points; the intent was to look at whether delivering the intervention affected the peer supporters' own reported behaviors as exploratory only. There was and is no intention to compare coach data to primary, secondary, or any other outcome measures of the randomized participants in the trial.

During the trial, another primary care center within the University of Michigan Health System was added. Because this center was within the University of Michigan Health System, and all contact information was identical, there was no reason to add another participating site.

ELIGIBILITY:
Inclusion Criteria:

Peer supporter:

* prior A1c 5.7 - 6.4 in last 3 years, with most recent being either lass than 5.7 or 0.4 points less than prior; AND/OR
* prior BMI >=25 or >=23 if Asian American in last three years with most recent 2% lower body weight;AND/OR
* prior completion of a wellness or diabetes prevention program; AND/OR
* completion of initial 6 months of UPSTART intervention as participant.

Patient participant:

* no prior dx of DM or current use of anti-hyperglycemic medication;
* BMI >=25 m2/kg or >=23 if Asian; and
* A1c 5.7 - 6.4.

Exclusion Criteria:

* serious psychiatric disorder in past 24 months
* pregnant or planning pregnancy
* substance abuse in past 12 months
* diagnosis of dementia, bipolar, schizophrenia, personality disorder
* other serious concerns rendering possible development of diabetes unimportant to potential participant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Elllen M Heisler, MD, Principal Investigator — University of Michigan; Julie A Schmittdiel, PhD, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente Northern California, Oakland, California
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heisler M, Dyer WT, Finertie H, Stoll SC, Wiley D, Turner CD, Sedgwick T, Kullgren J, Richardson CR, Hedderson M, Schmittdiel JA. Using Peer Support to Prevent Diabetes: Results of a Pragmatic RCT. Am J Prev Med. 2023 Aug;65(2):239-250. doi: 10.1016/j.amepre.2023.02.015. Epub 2023 Mar 8. PMID 36898949
- [Derived] Heisler M, Kullgren J, Richardson C, Stoll S, Alvarado Nieves C, Wiley D, Sedgwick T, Adams A, Hedderson M, Kim E, Rao M, Schmittdiel JA. Study protocol: Using peer support to aid in prevention and treatment in prediabetes (UPSTART). Contemp Clin Trials. 2020 Aug;95:106048. doi: 10.1016/j.cct.2020.106048. Epub 2020 Jun 1. PMID 32497783

RESULTS

PARTICIPANT FLOW:
Groups:
- Peer Support Arm (Intervention): Participants randomized to peer support will be matched with a peer supporter.
  Peer Support: Participants will be paired with a peer supporter. They will meet in person one time and then be in contact by phone or texting on a weekly basis for the first 6 months of a year.
  During the final six months of the year, the peer supporter and participant will be in touch at least monthly. The peer supporter will help link participants to existing health system and community diabetes prevention programs, support their engagement in formal programs, maintain achieved gains, and support participants to initiate and sustain healthy behaviors to prevent diabetes.
- Enhanced Usual Care (Control): Participants randomized to enhanced usual care will receive brief education and folder of information and resources.
  Enhanced Usual Care: Participants will receive brief education and folder of information and resources.
Period: Overall Study
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Started | 272 | 178
6-month Follow-up | 223 | 169
12-month Follow-up | 212 | 162
Completed | 219 | 162
Not Completed | 53 | 16
Not completed — Withdrawal by Subject | 53 | 16

BASELINE CHARACTERISTICS:
Population: Includes 95 peer supporters who delivered the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control) | Total
Number analyzed (Participants) | 272 | 178 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographics are presented separately by participant type: by the participants who were randomized and by the peer supporters who delivered the intervention.
  years
    Randomized Participants: number analyzed (Participants) | 177 | 178 | 355
    Randomized Participants | 55.8 (13.0) | 54.4 (12.9) | 55.1 (13.0)
    Peer Supporters: number analyzed (Participants) | 95 | 0 | 95
    Peer Supporters | 52.9 (14.1) |  | 52.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographics are presented separately by participant type: by the participants who were randomized and by the peer supporters who delivered the intervention.
  Participants
    Randomized Participants: number analyzed (Participants) | 177 | 178 | 355
    Randomized Participants: Female | 105 | 116 | 221
    Randomized Participants: Male | 72 | 62 | 134
    Peer Supporters: number analyzed (Participants) | 95 | 0 | 95
    Peer Supporters: Female | 64 |  | 64
    Peer Supporters: Male | 31 |  | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Demographics are presented separately by participant type: by the participants who were randomized and by the peer supporters who delivered the intervention.
  Participants
    Randomized Participants: number analyzed (Participants) | 177 | 178 | 355
    Randomized Participants: African American | 61 | 60 | 121
    Randomized Participants: Asian/Hawaiian Islander/Pacific Islander | 14 | 17 | 31
    Randomized Participants: Hispanic | 17 | 15 | 32
    Randomized Participants: Multiracial/Other | 11 | 15 | 26
    Randomized Participants: White | 74 | 71 | 145
    Peer Supporters: number analyzed (Participants) | 95 | 0 | 95
    Peer Supporters: African American | 32 |  | 32
    Peer Supporters: Asian/Hawaiian Islander/Pacific Islander | 11 |  | 11
    Peer Supporters: Hispanic | 7 |  | 7
    Peer Supporters: Multiracial/Other | 10 |  | 10
    Peer Supporters: White | 35 |  | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Randomized Participants | 177 | 178 | 355
  United States: Peer Supporters | 95 | 0 | 95
Highest Education Level [Count of Participants; unit: Participants] — Population: Demographics are presented separately by participant type: by the participants who were randomized and by the peer supporters who delivered the intervention.
  Participants
    Randomized Participant: number analyzed (Participants) | 177 | 178 | 355
    Randomized Participant: High School or Less / missing | 27 | 35 | 62
    Randomized Participant: College 1-3 years | 53 | 47 | 100
    Randomized Participant: College 4 or more years | 97 | 96 | 193
    Peer Supporters: number analyzed (Participants) | 95 | 0 | 95
    Peer Supporters: High School or Less / missing | 13 |  | 13
    Peer Supporters: College 1-3 years | 25 |  | 25
    Peer Supporters: College 4 or more years | 57 |  | 57
Annual Household Income [Count of Participants; unit: Participants] — Population: Demographics are presented separately by participant type: by the participants who were randomized and by the peer supporters who delivered the intervention.
  Participants
    Randomized Participant: number analyzed (Participants) | 177 | 178 | 355
    Randomized Participant: $0 - $30K | 43 | 33 | 76
    Randomized Participant: $31 - $55K | 24 | 32 | 56
    Randomized Participant: $56 - $100K | 39 | 44 | 83
    Randomized Participant: >$100K | 56 | 53 | 109
    Randomized Participant: Participant refused | 15 | 16 | 31
    Peer Supporter: number analyzed (Participants) | 95 | 0 | 95
    Peer Supporter: $0 - $30K | 19 |  | 19
    Peer Supporter: $31 - $55K | 21 |  | 21
    Peer Supporter: $56 - $100K | 18 |  | 18
    Peer Supporter: >$100K | 30 |  | 30
    Peer Supporter: Participant refused | 7 |  | 7
Self-Rated Health [Count of Participants; unit: Participants] — Data represents participants who self-rated their health as fair or poor. Population: Only participants randomized to this arm are included; peer supporters are not included.
  Participants
    number analyzed (Participants) | 177 | 178 | 355
    (all) | 33 | 36 | 69
Food Insecure [Count of Participants; unit: Participants] — Data represents participants who responded to the following statement with "Sometimes true" or "Often true": "We worried whether our food would run out before we got money to buy more." Population: Only participants randomized to this arm are included; peer supporters are not included.
  Participants
    number analyzed (Participants) | 177 | 178 | 355
    (all) | 26 | 33 | 59
Low Health Literacy [Count of Participants; unit: Participants] — Data represents participants who responded "Not at all", "A little", or "Somewhat" to the following question: "How confident are you filling out health care forms for yourself?" Population: Only participants randomized to this arm are included; peer supporters are not included.
  Participants
    number analyzed (Participants) | 177 | 178 | 355
    (all) | 20 | 19 | 39
Properties of Neighborhood [Mean (Standard Deviation); unit: units on a scale] — Properties of Neighborhood Scales take the average of responses (1 [strongly agree] to 5 [strongly disagree]) to a series of 7 questions used to assess neighborhood conditions that promote healthy behaviors, including walkability, access to gyms, availability of fruits and vegetables, and safety. This score ranges from 1 (neighborhood does not promote healthy behaviors or eating habits) to 5 (neighborhood promotes healthy behaviors and eating habits). Population: Only participants randomized to this arm are included; peer supporters are not included.
  units on a scale
    number analyzed (Participants) | 177 | 178 | 355
    (all) | 4.1 (0.8) | 4.1 (0.7) | 4.1 (0.8)
Major Depressive Disorder Likely [Count of Participants; unit: Participants] — Data represents participants where major depressive disorder is likely. PHQ-2 is a series of 2 questions used to screen for depression. Participants with a score between 3-6 (Major Depressive Disorder Likely) are represented here. Population: Only participants randomized to this arm are included; peer supporters are not included.
  Participants
    number analyzed (Participants) | 177 | 178 | 355
    (all) | 23 | 26 | 49
Glycosylated Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage] — An A1C test measures the percentage of red blood cells that have glucose-coated hemoglobin. This percentage indicates average blood sugar levels over the last 2-3 months. Higher percentages indicate higher levels of blood sugar levels, and an A1c between 5.7% and 6.4% is considered in the prediabetes range. Population: Only participants randomized to this arm are included; peer supporters are not included.
  Percentage
    number analyzed (Participants) | 177 | 178 | 355
    (all) | 5.9 (0.2) | 5.9 (0.2) | 5.9 (0.2)
Body Weight [Mean (Standard Deviation); unit: Kilograms] — Population: Only participants randomized to this arm are included; peer supporters are not included.
  Kilograms
    number analyzed (Participants) | 177 | 178 | 355
    (all) | 97.0 (21.9) | 97.1 (24.7) | 97.0371831 (23.3490493)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin A1c (HbA1c) at 6 Months
Description: An A1C test measures the percentage of red blood cells that have glucose-coated hemoglobin. This percentage indicates average blood sugar levels over the last 2-3 months. Higher percentages indicate higher levels of blood sugar levels, and an A1c between 5.7% and 6.4% is considered in the prediabetes range. The negative numbers for change over time indicate an improvement because they show a drop in percentages from the baseline percentages.
Time Frame: baseline to 6 months
Population: Data was unavailable for 23 participants in the Intervention arm and 37 participants in the Control arm because of scheduling issues and COVID.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 135 | 132
Percentage | -0.07 (0.20) | -0.06 (0.22)
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Outcomes were analyzed using multilevel models adapted for partially clustered data. Analyses was done in SAS v9.4; Test type: Superiority; p = 0.7436, Mixed Models Analysis

2. Primary Outcome: Change in Body Weight at 6 Months
Description: body weight in kilograms
Time Frame: baseline to 6 months
Population: Data was unavailable for 22 participants in the Intervention arm and 35 participants in the Control arm because of scheduling issues and COVID.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 136 | 134
Kilograms | -1.59 (4.76) | -0.70 (4.21)
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Outcomes were analyzed using multilevel models adapted for partially clustered data. Analyses was done in SAS v9.4; Test type: Superiority; p = 0.1212, Mixed Models Analysis

3. Secondary Outcome: Change in Glycosylated Hemoglobin A1c (HbA1c) at 12 Months
Description: as for outcome 1
Time Frame: baseline through 12 months
Population: Data was unavailable for 14 participants in the Intervention arm and 29 participants in the Control arm because of scheduling issues and COVID.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 137 | 133
Percentage | -0.06 (0.24) | -0.06 (0.27)
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Outcomes were analyzed using multilevel models adapted for partially clustered data. Analyses was done in SAS v9.4; Test type: Superiority; p = 0.8839, Mixed Models Analysis

4. Secondary Outcome: Change in Body Weight at 12 Months
Description: body weight in kilograms
Time Frame: baseline through 12 months
Population: Data was unavailable for 8 participants in the Intervention arm and 19 participants in the Control arm because of scheduling issues and COVID.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 143 | 143
Kilograms | -0.79 (5.99) | 0.22 (4.64)
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Outcomes were analyzed using multilevel models adapted for partially clustered data. Analyses was done in SAS v9.4; Test type: Superiority; p = 0.1137, Mixed Models Analysis

5. Secondary Outcome: Change in Whether Participant Enrolled in a Formal Program to Prevent Diabetes
Description: one item with yes/no response. Results indicate percentage of participants who responded "yes."
Time Frame: baseline through 12 months
Population: This measure only includes participants who, at baseline, had not enrolled in a formal program to prevent diabetes, and who answered the 12-month survey. For this reason, data was unavailable for 17 participants in the Intervention arm and 22 participants in the Control arm.
Measure: Number; unit: percentage of participants
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 134 | 140
percentage of participants | 25 | 14
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Outcomes were analyzed using multilevel models adapted for partially clustered data. Analyses was done in SAS v9.4; Test type: Superiority; p = 0.0162, Mixed Models Analysis

6. Secondary Outcome: Change in Number of Sessions Participant Attended in a Formal Program to Prevent Diabetes
Description: one item that asks participant to report number of sessions attended
Time Frame: baseline through 12 months
Population: Measure was initially conceived of as a face-to-face session. However, when the trial began, additional sessions became available online because of COVID and an increase in online offerings. As a result, no data was collected for this measure.
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Frequency and Duration Participant Engages in Moderate to Vigorous Physical Activity as Shown by Minutes Per Week
Description: This combined measure is based on participant-reported frequency and duration of moderate to vigorous physical activity, measured in minutes per week. Frequency and duration were initially registered separately.
  Two questions were used to calculated minutes of physical activity per week, asked in both the baseline and 12 months surveys:
  Q1. On average, how many days per week do you engage in moderate-to-vigorous physical activity? A1: 0-7, integer response only Q2: On average on those days, how many minutes do you engage in physical activity as this level? A2: open numeric response
  A1*A2 = minutes per week (Physical Activity value)
  Minutes of physical activity per week reported in 12 month survey - minutes of physical activity per week in baseline survey = change in minutes per week of physical activity
Time Frame: baseline through 12 months
Population: Survey responses/data were unavailable for 20 participants from the Intervention arm and 22 from the Control arm because some participants never completed either a baseline or a 12-month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 131 | 140
Minutes | 30.00 [-40.00 to 105.00] | 7.50 [-30.00 to 75.00]
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Outcomes were analyzed using multilevel models adapted for partially clustered data. Analyses was done in SAS v9.4; Test type: Superiority; p = 0.2117, Mixed Models Analysis

8. Secondary Outcome: Change in the Number of Times Drinking Regular Soda or Pop That Contains Sugar
Description: Recorded frequency of consumption in the last 30 days. Participants could report times per day, times per week, or times over past 30 days. These reports were converted to the number of times over past 30 days participants drank regular soda or pop that contained sugar.
Time Frame: baseline through 12 months
Population: Survey responses/data were unavailable for 20 participants from the Intervention arm and 23 from the Control arm because some participants never completed either a baseline or a 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded.
Measure: Median (Inter-Quartile Range); unit: Times Consumed
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 131 | 139
Times Consumed | 0.00 [-3.00 to 0.00] | 0.00 [-1.00 to 0.00]
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Superiority; p = 0.4169, Mixed Models Analysis

9. Secondary Outcome: Change in Patient Activation as Measured by the Patient Activation Measure 13 (PAM-13)
Description: PAM-13 is a 13-item scale that measures participant beliefs, perceived knowledge, and confidence for engaging in behaviors related to the participant's health condition. PAM-13 has a 0-100 scale, where a low score indicates low activation (disengaged and overwhelmed) and a high score indicates high activation (patient considers self their own advocate). The difference between the score at 12 months and the score at baseline was calculated.
Time Frame: baseline through 12 months
Population: Survey responses/data were unavailable for 17 participants from the Intervention arm and 23 from the Control arm because some participants never completed either a baseline or a 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 134 | 139
units on a scale | 1.12 (13.34) | 1.80 (14.13)
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Outcomes were analyzed using multilevel models adapted for partially clustered data. Analyses was done in SAS v9.4; Test type: Superiority; p = 0.8785, Mixed Models Analysis

10. Secondary Outcome: Change in Participant's Perceived Confidence in Their Ability to Take Steps to Prevent Diabetes Using the Williams Perceived Competence Scale
Description: Williams Perceived Competence Scale comprises 4 items measuring the participants' perception of their own ability to take steps to prevent diabetes. Responses for each individual question range from 1 (not at all true) to 7 (very true). The responses to all 4 items were averaged (range: 1-7), with higher scores on the scale indicating higher perceived competence in preventing diabetes.
Time Frame: baseline through 12 months
Population: Survey responses/data were unavailable for 18 participants from the Intervention arm and 22 from the Control arm because some participants never completed either a baseline or a 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 133 | 140
units on a scale | -0.34 (1.32) | -0.52 (1.26)
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Outcomes were analyzed using multilevel models adapted for partially clustered data. Analyses was done in SAS v9.4; Test type: Superiority; p = 0.1006, Mixed Models Analysis

11. Secondary Outcome: Change in Autonomous Motivation to Prevent Diabetes Using the Treatment Self-Regulation Questionnaire (TSRQ - Autonomous)
Description: The Treatment Self-Regulation Questionnaire (TSRQ) consisted of 11 items that measured the participants' perceptions of how true various reasons to take steps to help prevent diabetes may be to the participants.
  The TSRQ was split into two measures: autonomous and controlled. The autonomous measure consisted of 4 items that measured participants' autonomous (or internal) perceptions of how true various reasons to take steps to help prevent diabetes may be to the participants.
  Responses for each individual question range from 1 (not at all true) to 7 (very true). The responses to all 4-items are averaged (range: 1-7). Higher scores indicate participants agree with more internal reasons for preventing diabetes (ex: wanting to take responsibility for my own health).
Time Frame: baseline through 12 months
Population: Survey responses/data were unavailable for 18 participants from the Intervention arm and 23 from the Control arm because some participants never completed either a baseline or a 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded.
Measure: Mean (Standard Deviation); unit: score on a questionnaire
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 133 | 139
score on a questionnaire | -0.06 (0.60) | -0.05 (0.68)
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Superiority; p = 0.7168, Mixed Models Analysis

12. Secondary Outcome: Change in the Participant's Level of Social Support Related to Improving Their Own Health Behaviors Using the Change in Health-Specific Social Support Scale
Description: The Health-Specific Social Support Scale consisted of 12 items that asked participants to indicate their level of agreement on a 6-point Likert scale ("Strongly disagree" [1] to "Strongly agree" [6]) with statements regarding accessibility of any contact they had with people in the past 3 months who were specifically also at risk for developing diabetes and could provide social support in attempts to prevent diabetes via healthy lifestyle changes. Scores for negative statements were reversed, and the total score was the sum of all scores. Total scores can range from 12 (minimum) to 72 (maximum). A higher score indicated a better outcome because it indicated a higher level of reported social support.
Time Frame: baseline through 12 months
Population: Survey responses/data were unavailable for 22 participants from the Intervention arm and 26 from the Control arm because some participants never completed either a baseline or a 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 129 | 136
units on a scale | 9.34 (12.13) | 3.69 (13.59)
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Outcomes were analyzed using multilevel models adapted for partially clustered data. Analyses was done in SAS v9.4; Test type: Superiority; p = 0.0001, Mixed Models Analysis

13. Secondary Outcome: The Role a Participant's Peer Supporter Played in Assisting Them to Set and Reach Their Goals Using the Goal Setting and Intervention Tailoring Subscale of the Patient Assessment of Chronic Illness Care (PACIC) at 6 Months
Description: The goal setting and intervention tailoring subscale of the Patient Assessment of Chronic Illness Care (PACIC) consisted of 5 questions that ask the participant to state how often their peer supporter engaged in supportive behaviors regarding setting and achieving goals in order to make healthy lifestyle changes. Each question had a range of 1 (None of the time) to 5 (Always). Averaged scores range from 1 (minimum) to 5 (maximum). A higher score indicated a better outcome because it indicated that the peer perceived their partner to be more supportive.
Time Frame: 6 months
Population: Survey responses/data were unavailable for 20 participants from Intervention arm because some participants never completed a baseline or 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded. For these specific intervention-only questions, some peers were never assigned a coach and therefore skipped these questions regarding coach interactions. Participants in the Enhanced Usual Care (Control) arm were not assigned a peer supporter.
Measure: Mean (Standard Deviation); unit: Score on a questionnaire
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 138 | 0
Score on a questionnaire | 3.79 (0.89) |
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Other — Single group analysis for peer support group only; Mean = 3.799, Standard Deviation 0.885

14. Secondary Outcome: The Role a Participant's Peer Supporter Played in Assisting Them to Set and Reach Their Goals Using the Goal Setting and Intervention Tailoring Subscale of the Patient Assessment of Chronic Illness Care (PACIC) at 12 Months
Description: as for outcome 13
Time Frame: 12 months
Population: Survey responses/data were unavailable for 27 participants from Intervention arm because some participants never completed a baseline or 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded. For these specific intervention-only questions, some peers were never assigned a coach and therefore skipped these questions regarding coach interactions. Participants in the Enhanced Usual Care (Control) arm were not assigned a peer supporter.
Measure: Mean (Standard Deviation); unit: Score on a questionnaire
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 124 | 0
Score on a questionnaire | 3.73 (0.99) |
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Other — Single group analysis for peer support group only; Mean = 3.732, Standard Deviation 0.985

15. Secondary Outcome: Participant's Perceived Autonomy Support From Their Peer Supporter Using the Health Care Climate Questionnaire (HCCQ, Long Form) at 6 Months
Description: The Health Care Climate Questionnaire (HCCQ, long form) consisted of 15 items that asked the participant to rank their agreement with statements that indicated degree of autonomy support (Strongly Disagree [1] to Strongly Agree [7]). Averaged scores ranged from 1 (minimum) to 7 (maximum). A higher the score indicated a better outcome because it indicated that the peer perceived their partner to be more autonomy supportive.
Time Frame: 6 months
Population: Survey responses/data were unavailable for 20 participants from the Intervention arm because some participants never completed a baseline or 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded. For these specific intervention-only questions, some peers were never assigned a coach and therefore skipped these questions regarding coach interactions. Participants in the Enhanced Usual Care (Control) arm were not assigned a peer supporter.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 138 | 0
score on a scale | 6.22 (1.08) |
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Other — Single group analysis for peer support group only; Mean = 6.222, Standard Deviation 1.083

16. Secondary Outcome: Participant's Perceived Autonomy Support From Their Peer Supporter Using the Health Care Climate Questionnaire (HCCQ, Long Form) at 12 Months
Description: The Health Care Climate Questionnaire (HCCQ, long form) consisted of 15 items that asked the participants to rank their agreement with statements that indicated degree of autonomy support (Strongly Disagree [1] to Strongly Agree [7]). Total scores ranged from 1 (minimum) to 7 (maximum). A higher score indicated a better outcome because it indicated that the peer perceived their partner to be more autonomy supportive.
Time Frame: 12 months
Population: Survey responses/data were unavailable for 27 participants from the Intervention arm because some participants never completed a baseline or 12-month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded. For these specific intervention-only questions, some peers were never assigned a coach and therefore skipped these questions regarding coach interactions. Participants in the Enhanced Usual Care (Control) arm were not assigned a peer supporter.
Measure: Mean (Standard Deviation); unit: Score on Questionnaire
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 124 | 0
Score on Questionnaire | 6.18 (1.14) |
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Other — Single group analysis for peer support group only; Mean = 6.179, Standard Deviation 1.141

17. Secondary Outcome: Change in the Number of Times Drinking Sugary Drinks Besides Pop or Soda
Description: Recorded frequency of consumption in the last 30 days. Participants could report times per day, times per week, or times over past 30 days. These reports were converted to the number of times over past 30 days participants drank sugary drinks besides pop or soda.
Time Frame: baseline through 12 months
Population: Survey responses/data were unavailable for 19 participants from the Intervention arm and 24 from the Control arm because some participants never completed either a baseline or a 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded.
Measure: Median (Inter-Quartile Range); unit: Times Consumed
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 132 | 138
Times Consumed | 0.00 [-5.00 to 0.00] | 0.00 [-4.30 to 2.00]
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Superiority; p = 0.9126, Mixed Models Analysis

18. Secondary Outcome: Change in the Number of Times Eating Fruit
Description: Recorded frequency of consumption in the last 30 days - participants could report times per day, times per week, or times over past 30 days, which was converted to times over past 30 days
Time Frame: baseline through 12 months
Population: Survey responses/data were unavailable for 19 participants from the Intervention arm and 22 from the Control arm because some participants never completed either a baseline or a 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded.
Measure: Median (Inter-Quartile Range); unit: Times Consumed
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 132 | 140
Times Consumed | 0.00 [-10.60 to 8.60] | 0.00 [-8.50 to 7.55]
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Superiority; p = 0.7405, Mixed Models Analysis

19. Secondary Outcome: Change in the Number of Times Eating Vegetables
Description: One measure that recorded frequency of consumption in the last 30 days - participants could report times per day, times per week, or times over past 30 days, which was converted to times over past 30 days
Time Frame: baseline through 12 months
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Times Consumed
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 133 | 140
Times Consumed | 0.00 [-4.30 to 8.60] | 0.00 [-12.80 to 12.90]
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Superiority; p = 0.5956, Mixed Models Analysis

20. Secondary Outcome: Change in the Number of Times Eating Meals Cooked With Olive Oil
Description: as for outcome 19
Time Frame: baseline through 12 months
Population: Survey responses/data were unavailable for 19 participants from the intervention arm and 23 from the control arm because some participants never completed either a baseline or a 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded.
Measure: Median (Inter-Quartile Range); unit: Times Consumed
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 132 | 139
Times Consumed | 0.00 [-4.30 to 7.50] | 0.00 [-6.60 to 8.60]
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Superiority; p = 0.3341, Mixed Models Analysis

21. Secondary Outcome: Change in the Number of Times Eating Sweets or Desserts
Description: as for outcome 19
Time Frame: baseline through 12 months
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Times Consumed
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 133 | 140
Times Consumed | -3.60 [-9.00 to 0.30] | -4.30 [-16.30 to 4.30]
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Superiority; p = 0.2049, Mixed Models Analysis

22. Secondary Outcome: Change in the Number of Times Eating Whole Grain Breads, Whole Grain Pasta, or Brown Rice
Description: as for outcome 19
Time Frame: baseline through 12 months
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Times Consumed
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 133 | 140
Times Consumed | 0.00 [-7.60 to 8.60] | 0.00 [-9.25 to 4.80]
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Superiority; p = 0.0335, Mixed Models Analysis

23. Secondary Outcome: Change in the Number of Times Eating Breads, Pasta, Rolls, or Rice Made From White, Refined Grains
Description: as for outcome 19
Time Frame: baseline through 12 months
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: Times Consumed
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 132 | 140
Times Consumed | -0.15 [-6.60 to 3.00] | 0.00 [-8.60 to 4.10]
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Superiority; p = 0.3219, Mixed Models Analysis

24. Secondary Outcome: Change in Controlled Motivation to Prevent Diabetes Using the Treatment Self-Regulation Questionnaire (TSRQ - Controlled)
Description: The Treatment Self-Regulation Questionnaire (TSRQ) consists of 11 items that measure participants' perceptions of how true various reasons to take steps to help prevent diabetes may be to the participants.
  The TSRQ is split into two measures: autonomous and controlled. The controlled measure consists of 7 items that measure participants' controlled (or external) perceptions of how true various reasons to take steps to help prevent diabetes may be to the participants.
  Responses for each individual question range from 1 (not at all true) to 7 (very true). The responses to all 7-items are averaged (range: 1-7). Higher scores indicate participants agree with more external behaviors or reasons for preventing diabetes (ex: feeling pressure to do so from others).
Time Frame: baseline through 12 months
Population: Survey responses/data were unavailable for 20 participants from the intervention arm and 26 from the control arm because some participants never completed either a baseline or a 12 month survey. Additionally, KPNC allowed participants to skip survey questions, so some may not have responded.
Measure: Mean (Standard Deviation); unit: score on a questionnaire
Arm/Group | Peer Support Arm (Intervention) | Enhanced Usual Care (Control)
Number analyzed (Participants) | 131 | 136
score on a questionnaire | 0.07 (1.09) | 0.20 (1.16)
Statistical Analysis 1: Comparison: Peer Support Arm (Intervention) vs Enhanced Usual Care (Control); Test type: Superiority; p = 0.5223, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 12 months for each participant
Arm/Group | Enhanced Usual Care (Control) | Peer Support Arm (Intervention)
All-Cause Mortality (participants affected / at risk) | 0/178 | 1/177
Serious Adverse Events (participants affected / at risk) | 0/178 | 0/177
Other Adverse Events (participants affected / at risk) | 0/178 | 0/177

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT03689530/Prot_SAP_000.pdf